CLINICAL TRIAL: NCT00300105
Title: A Parallel-Group, Multi-Centre, Active-Controlled (Glibenclamide) Long-Term Extension Study to Evaluate the Safety and Tolerability of Oral Tesaglitazar Therapy in Patients With Type 2 Diabetes
Brief Title: GALLEX 4 - Long-Term Extension Study to Evaluate Tesaglitazar Therapy in Patients With Type 2 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The development program has been terminated
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6160C00047; EudraCT No 2004-005243-97
Record Dates: First submitted 2006-03-07; First posted 2006-03-08 (Estimated); Last update posted 2008-03-17 (Estimated); Status verified 2008-03

CONDITIONS: Type 2 Diabetes
Keywords: Patients diagnosed with type 2 diabetes who have participated in and completed the randomized, double-blind, parallel-group, multi-center study GALLANT 4
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — tesaglitazar

INTERVENTIONS:
Drug: Tesaglitazar

SUMMARY:
This is a parallel-group, multi-center, long-term extension study from the GALLANT 4 study to monitor the safety and tolerability of oral tesaglitazar compared with glibenclamide in patients with type 2 diabetes for up to 100 weeks of treatment. The total duration, including treatment and follow-up, is 103 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a written informed consent
* Men or women who are >=18 years of age
* Female patients: postmenopausal, hysterectomized, or if of childbearing potential, using a reliable method of birth control
* Completed the last two visits of randomized treatment period in GALLANT 4

Exclusion Criteria:

* Type 1 diabetes
* New York Heart Association heart failure Class III or IV
* Treatment with chronic insulin
* History of hypersensitivity or intolerance to any peroxisome proliferator-activated receptor agonist (like Actos or Avandia), fenofibrate, metformin or 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitor (statin)
* History of drug-induced myopathy or drug-induced creatine kinase elevation, liver enzyme elevations, neutropenia (low white blood cells)
* Creatinine levels above twice the normal range
* Creatine kinase above 3 times the upper limit of normal
* Previous enrollment in this long-term extension study
* Any clinically significant abnormality identified on physical examination, laboratory tests or electrocardiogram, which in the judgment of the investigator would compromise the patient's safety or successful participation in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2005-10; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Adverse events, laboratory variables, physical examination, cardiac evaluation, hypoglycemic events, electrocardiogram, vital signs (blood pressure and pulse), body weight

SECONDARY OUTCOMES:
Effect of tesaglitazar versus glibenclamide, with or without other oral anti-diabetic drugs on
Time to treatment failure
Changes in glycemic variables: glycosylated hemoglobin A1c and fasting plasma glucose (FPG)
Responder rates and proportion of patients who reach pre-specified target levels for glycosylated hemoglobin A1c and FPG
Markers of insulin resistance by assessment of insulin homeostasis assessment model
Preventing beta-cell function by assessment of changes in the ratios proinsulin/insulin and C-peptide/FPG
Changes in lipid variables (triglyceride, total cholesterol, high-density lipoprotein cholesterol [HDL-C], non-HDL-C, low-density lipoprotein cholesterol, low-density lipoprotein cholesterol/HDL-C, apolipoprotein [Apo] B, ApoA-1, ApoB/ApoA-1
Responder rates and proportion of patients who reach pre-specified target levels for triglyceride and HDL-C
Inflammatory and coagulability markers by assessment of C-reactive protein, fibrinogen, tumor necrosis factor-alpha, and intracellular adhesion molecule-1
Urinary albumin excretion
Central obesity (waist circumference, hip circumference and waist/hip ratio)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Galida Medical Science Director, MD, Study Director — AstraZeneca
Locations (42):
- Belgium (4):
  - Research Site, Hasselt
  - Research Site, Liège
  - Research Site, Sint-Gillis-Waas
  - Research Site, Steenokkerzeel
- Research Site, Shatin, Hong Kong
- Hungary (5):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Székesfehérvár
- Italy (6):
  - Research Site, Gubbio
  - Research Site, Milan
  - Research Site, Perugia
  - Research Site, Piacenza
  - Research Site, Reggio Emilia
  - Research Site, Udine
- Malaysia (2):
  - Research Site, Kubang Kerian, Kelantan
  - Research Site, Kuala Lumpur
- Philippines (3):
  - Research Site, Makati City
  - Research Site, Manila
  - Research Site, Pasig
- Poland (7):
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Płock
  - Research Site, Torun
  - Research Site, Tychy
  - Research Site, Warsaw
  - Research Site, £ód?
- Slovakia (10):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Ilava
  - Research Site, Košice
  - Research Site, Kysucké Nové Mesto
  - Research Site, Lučenec
  - Research Site, Ľubochňa
  - Research Site, Nitra
  - Research Site, Prešov
  - Research Site, Trnava
- South Africa (3):
  - Research Site, Johannesburg, Gauteng
  - Research Site, Cape Town
  - Research Site, Durban
- Research Site, Bangkok, Thailand